CLINICAL TRIAL: NCT04361370
Title: A Single-arm Phase II Study of Olaparib Maintenance With Pembrolizumab & Bevacizumab in BRCA Non-mutated Patients With Platinum-sensitive Recurrent Ovarian Cancer (OPEB-01)
Brief Title: Olaparib Maintenance With Pembrolizumab & Bevacizumab in BRCA Non-mutated Patients With Platinum-sensitive Recurrent Ovarian Cancer
Acronym: OPEB-01
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0386
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Platinum-sensitive Recurrent BRCA Wild Type Ovarian Cancer
Keywords: BRCA wild type; ovarian cancer; Platinum-sensitive
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): BRCA mutation wild type, non-mucinous , platinum-sensitive recurrent ovarian cancer
  Interventions: Drug: Olaparib-Pembrolizumab-Bevacizumab

INTERVENTIONS:
Drug: Olaparib-Pembrolizumab-Bevacizumab — * Olaparib 300mg (twice daily [BID])
  * Pembrolizumab 200mg every 3 weeks (Q3W) from 2nd infusion for up to 35 infusions
  * Bevacizumab 15mg/kg or 7.5mg/kg every 3 weeks (Q3W)

SUMMARY:
This study is phase II, open label, clinical trial to determine the efficacy of Olaparib maintenance with Bevacizumab and Pembrolizumab by assessment progression-free survival(6 months PFS rate) in BRCA non-mutated patients with platinum-sensitive recurrent ovarian cancer.

DETAILED DESCRIPTION:
'This is a Phase II, open-label, non-randomized, multi-center study assessing the efficacy and safety of Olaparib maintenance with Bevacizumab and Pembrolizumab in subjects with platinum-sensitive who have received prior of platinum-based chemotherapy. The study will assess the effectiveness of progression-free survival(6 months PFS rate) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The subject will be treated to until disease progression as below:

* Maintenance : Olaparib 300mg (twice daily [BID])
* Pembrolizumab 200mg every 3 weeks (Q3W) from 2nd infusion for up to 35 infusions
* Bevacizumab 15mg/kg or 7.5mg/kg every 3 weeks (Q3W)

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed diagnosis of high-grade predominantly serous, endometrioid, carcinosarcoma, mixed mullerian with high-grade serous component, clear cell, or low-grade serous OC, primary peritoneal cancer, or fallopian tube cancer will be enrolled in this study (only up to 8 patients with clear cell carcinoma will be included and mucinous carcinoma will not be included).
* Participant has received 2 previous courses of platinum-containing therapy, and has disease that was considered platinum sensitive following the penultimate (next to last) platinum course (more than 6 months' period between penultimate platinum regimen and progression of disease
* Participant has responded to last the platinum regimen (complete or partial response), remains in response and is enrolled on study within 8 weeks of completion of the last platinum regimen
* Participant is able to provide a newly obtained core or excisional biopsy of a tumor lesion for prospective testing of BRCA 1/2 and PD-L1 status prior to enrollment
* Female participants who are at least 20 years of age and Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participant has adequate organ function as defined in the following:

  1. ANC≥1500/µL
  2. PLT≥100 000/µL
  3. Hemoglobin≥9.0 g/dL or ≥5.6 mmol/L
  4. Creatinine≤1.5 × ULN or calculated creatinine clearance≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
  5. Total bilirubin≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
  6. AST (SGOT) and ALT (SGPT)≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
  7. International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT)≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Participant has mucinous, germ cell, or borderline tumor of the ovary
* Participant has a known or suspected deleterious mutation (germline or somatic) in either BRCA1 or BRCA2
* Participant has a history of non-infectious pneumonitis that required treatment with steroids or currently has pneumonitis
* Participant either has myelodysplastic syndrome (MDS)/ acute myeloid leukemia (AML) or has features suggestive of MDS/AML
* Participant has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Participant has known active CNS metastases and/or carcinomatous meningitis
* Participant has a known history of active TB (Bacillus Tuberculosis)
* Participant has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
* Participant has uncontrolled hypertension, defined as systolic > 140 mmHg or diastolic > 90 mmHg documented by 2 blood pressure readings taken at least 1 hour apart
* Participant has a history of hemorrhage, hemoptysis or active gastrointestinal bleeding within 6 months prior to randomization

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(6 months PFS rate) | 6 months
  To determine the clinical effectiveness of the study treatment assessed using progression free survival(6months) according to RECIST v1.1 criteria (Investigator determined)

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 1year
Time to tumour progression (TTP) | Up to 1year
Time to first subsequent treatment(or death) | The date of first documented first subsequent treatment or date of death, assessed up to 72 months
Time to second subsequent treatment | The date of first documented second subsequent treatment assessed up to 72 months
progression-free survival | Up to 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YJ, Lim MC, Kim BG, Ngoi NY, Choi CH, Park SY, Tan DS, Go Y, Lee JY. A single-arm phase II study of olaparib maintenance with pembrolizumab and bevacizumab in BRCA non-mutated patients with platinum-sensitive recurrent ovarian cancer (OPEB-01). J Gynecol Oncol. 2021 Mar;32(2):e31. doi: 10.3802/jgo.2021.32.e31. Epub 2021 Jan 27. PMID 33559413